CLINICAL TRIAL: NCT04993742
Title: Effects of Pregnancy-Specific Anxiety on Placental Inflammatory and Oxidative Stress Response and Birth Outcomes (MOMS Placenta)
Brief Title: Effects of Pregnancy-Specific Anxiety on Placental Inflammatory and Oxidative Stress Response and Birth Outcomes
Acronym: MOMSPlacenta
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: 59th Medical Wing (U.S. Federal Agency); Brooke Army Medical Center (U.S. Federal Agency); University of the Incarnate Word (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FWH20190163H
Record Dates: First submitted 2020-11-02; First posted 2021-08-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Placental Dysfunction; Prenatal Stress
Keywords: placenta; prenatal; pregnancy; maternal anxiety; prenatal depression; biomarker

STUDY DESIGN:
Intervention Model Description: The study is a repeated measures, longitudinal design
Masking Description: Coded histopathology slides will be sent to pathologist for evaluation with only a study number
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOMS Intervention (Experimental): Women that are currently in the Mentors Offering Maternal Support (M-O-M-S) research program as well as pregnant women entering prenatal care in the first trimester, who are not in the M-O-M-S program may participate in the study.
  Arms Assigned Interventions Experimental: M-O-M-S Intervention M-O-M-S intervention is 10, 1 hour prenatal mentored support groups
  No Intervention: Routine Prenatal Care Routine prenatal care in accordance with the Department of Defense Pregnancy Guidelines
  Interventions: Behavioral: MOMS Intervention

INTERVENTIONS:
Behavioral: MOMS Intervention — Behavioral: Mentors Offering Maternal Support (M-O-M-S) 10, 1 hour, structured classes meeting every-other-week in person beginning in the first trimester of pregnancy and unlimited access to mentor support.

SUMMARY:
Explore the associations of prenatal maternal anxiety to placental histologic findings, and the pro-inflammatory, anti-inflammatory, and immunoregulatory cells found in the placenta and determine the effect of maternal anxiety on the association between placental molecular changes on pregnancy and birth and infant outcomes.

DETAILED DESCRIPTION:
Purpose: Explore the associations of prenatal maternal anxiety to placental histologic findings, and the pro-inflammatory, anti-inflammatory, and immunoregulatory cells found in the placenta and determine the effect of maternal anxiety on the association between placental molecular changes on pregnancy and birth and infant outcomes.

Subject Population: Prenatal patients receiving obstetrical care at the Brooke Army Medical Center (BAMC) will be the focused population. Patients must be 18 years or older and planning to deliver at the BAMC.

Design: This study is a longitudinal prospective, randomized clinical trial with repeated measures of independent groups to investigate both psychosocial and physiologic data in the early prenatal, maternal intervention (Mentors Offering Maternal Support, M-O-M-S™), to standard prenatal care without the M-O-M-S, for decreasing maternal prenatal anxiety and depression, and reducing maternal inflammatory and oxidative stress responses.

Procedures: Participants will be randomized to the treatment arm (M-O-M-S™) or the control group (prenatal care without M-O-M-S™). Participants will complete multiple psychosocial measures questionnaires at initial recruitment and at approximately 16, 24, 28 and 32 weeks gestation. Women randomized to the M-O-M-S™ program will attend 10 sessions, lasting 1 hr. every-other-week.

Maternal whole peripheral blood collection will be performed in conjunction with the participant's normal prenatal blood draw at 4-10, 16-20, and 28-32 weeks gestation. At each datapoint, blood will be collected in one 2.5 ml serum separator tube. The serum separator vacutainer will be centrifuged, and the serum placed in aliquots per participant sample. Maternal serum collected will be analyzed to quantify Th1, Th2, and Th17 cytokine levels, and oxidative stress and hormonal biomarkers. The isolated serum samples will be frozen and transported to the 59MDW CIRS laboratory at JBSA Lackland for processing, aliquoting and storage. The samples will be stored in a repository at CIRS for future comprehensive-omics analysis.

Participant placentas delivered will be sent to SAMMC/BAMC pathology laboratory where the placental examination as recommended by the College of American Pathologists will be completed. Placental tissue biopsies will be collected, gross and microscopic examinations will occur. Histopathological findings will be classified according to standard guidelines and coded into categories that identify vascular malperfusion or uteroplacental vascular insufficiency, chorion regression syndrome, and other maternal inflammatory disorders. Dr. Brady (PI) and/or the pathology residents will conduct the initial examination and determine placental diagnosis, which will then be confirmed by another expert blinded to all clinical details in order to remove interpretative bias and establish interrater reliability. The placental tissue samples will also be used for proteomic analyses. Placental tissue biopsies, taken from the same locations as the tissue for the histological paraffin blocks, will be flash-frozen in liquid nitrogen.

Both the serum and placental tissues will be isolated and frozen prior to transport and sent (by courier) to the 59 MDW Clinical Investigations & Research Support (CIRS) Laboratory at JBSA-Lackland for processing, aliquoting, and storage. Serum and placental tissue samples will be stored in a repository at CIRS for future comprehensive -omics analyses.

ELIGIBILITY:
Inclusion Criteria:

* All Active Duty and DoD beneficiary gravid women,
* 18 years of age or older,
* Receiving prenatal care at BAMC,
* English speaking

Exclusion Criteria:

* Military dependent daughters
* VA beneficiaries

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Explore associations between prenatal maternal psychosocial measures of anxiety depression with immunological, oxidative stress, and hormonal biomarker changes found in maternal serum with and without the M-O-M-S™ support intervention. | at time of MOMS intervention administer
  Correlate % of participants with increased measures of anxiety and depression will be associated with changes in Th1, Th2, and Th17 responses as well as an increase in hormonal and oxidative stress biomarkers indicative of a proinflammatory and physiological stressed state.
Explore associations between prenatal maternal psychosocial measures of anxiety depression with immunological, oxidative stress, and hormonal biomarker changes found in placental tissue with and without the M-O-M-S™ pregnancy intervention. | at time of maternal serum and placental tissue collection
  Correlate % of participants with increased measures of anxiety and depression will be associated with changes in Th1, Th2, and Th17 responses as well as an increase in hormonal and oxidative stress biomarkers within the placental tissue indicative of a pro-inflammatory and physiological stressed state that is correlative to changes in maternal serum.
Explore associations between prenatal maternal psychosocial measures of anxiety and depression to histopathology changes in placental tissue with and without the M-O-M-S™ intervention. | at time of placental tissue collection
  Correlate% of participants with increased measures of pregnancy anxiety and depression will be associated with the development of maternal vascular malperfusion or uteroplacental vascular insufficiency, chorion regression syndrome, and maternal inflammatory disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Tony T Yuan, PhD, Principal Investigator — Uniformed Services University of the Health Sciences; Robert O Brady, MD, Principal Investigator — 59 Medical Wing; Karen L Weis, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Joint Base San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Result] Weis KL, Yuan TT, Walker KC, Gibbons TF, Chan W. Associations between Physiological Biomarkers and Psychosocial Measures of Pregnancy-Specific Anxiety and Depression with Support Intervention. Int J Environ Res Public Health. 2021 Jul 29;18(15):8043. doi: 10.3390/ijerph18158043. PMID 34360332
- [Result] Weis KL, Ryan TW. Mentors offering maternal support: a support intervention for military mothers. J Obstet Gynecol Neonatal Nurs. 2012 Mar;41(2):303-314. doi: 10.1111/j.1552-6909.2012.01346.x. PMID 22834852
- [Result] Weis KL, Lederman RP, Lilly AE, Schaffer J. The relationship of military imposed marital separations on maternal acceptance of pregnancy. Res Nurs Health. 2008 Jun;31(3):196-207. doi: 10.1002/nur.20248. PMID 18213640
- [Result] Weis KL, Lederman RP, Walker KC, Chan W. Mentors Offering Maternal Support Reduces Prenatal, Pregnancy-Specific Anxiety in a Sample of Military Women. J Obstet Gynecol Neonatal Nurs. 2017 Sep-Oct;46(5):669-685. doi: 10.1016/j.jogn.2017.07.003. Epub 2017 Jul 24. PMID 28751158

DOCUMENTS (2):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT04993742/Prot_000.pdf
  • Informed Consent Form (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT04993742/ICF_002.pdf